CLINICAL TRIAL: NCT00832468
Title: The Complementary Effect of Ear Acupressure on Older Patients With Chronic Insomnia and Anxiety
Brief Title: The Complementary Effect of Ear Acupressure on Older Patients With Chronic Insomnia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Yen-Ying Kung, Institute of Traditional Medicine, National Yang-Ming University, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 97032R
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Last update posted 2009-12-08 (Estimated); Status verified 2009-12

CONDITIONS: Insomnia
Keywords: insomnia; ear acupressure
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sham ear acupressure (Placebo Comparator)
  Interventions: Other: sham ear acupressure
- ear acupressure (Experimental)
  Interventions: Other: ear acupressure

INTERVENTIONS:
Other: ear acupressure — The ear acupressure that is used involved a 0.3 cm-sized magnetic pellet on a 1 cm size sticky patch (Ching-Ming Co., Taiwan), which was placed on the bilateral ear Shenmen points; each of the points were pressed once a second for one minute (60 times) before sleep every night. The time period of the treatment course was four weeks.
  Arms: ear acupressure
Other: sham ear acupressure — The sham ear acupressure that was used involved a 1 cm size sticky patch placed on the bilateral ear Shenmen points. There was no magnetic pellet attached to the sticker and no need to press it.
  Arms: sham ear acupressure

SUMMARY:
Ear acupressure is commonly applied to treat insomnia in Oriental clinical practice but lacking the evidence of the randomized controlled trial (RCT)of ear acupressure on insomnia. In this study, a RCT is conducted to investigate the complementary effect of ear acupressure on chronic insomnia in old adults.

DETAILED DESCRIPTION:
Even though there have been many advances in the pharmacological treatment of insomnia, many patients with insomnia visit complementary and alternative medicine (CAM) specialists for help due to fear of the side effects of long-term treatment with hypnotics. Acupuncture is commonly used to treat insomnia in the field of CAM. Among the different methods of acupuncture, it has been noted that ear acupressure (placing magnetic pellets on the auricular points), which has the advantage of being non-invasive and easily carried out, shows possible effects whereby there is improvement in the sleep quality of old adults. However, it is lacking of the evidence of the randomized controlled trial (RCT) of ear acupressure on insomnia.

Insomnia is related to homeostatic dysregulation of autonomic nervous system (ANS). Ear acupuncture and its related techniques are believed to act through the reticular formation and the ANS may thus result in an amelioration of illness.

In this study, a RCT is conducted to investigate the complementary effect of ear acupressure on chronic insomnia in old adults.Besides, the changes of ANS function (measured by heart rate variability) are recorded to evaluate the role of ANS in the treatment of insomnia.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of primary insomnia

Exclusion Criteria:

* diabetic neuropathy
* cardiac arrythmia
* liver disease (ALT> 120 U/L)
* renal disease (Cr> 2 mg/dl)
* severe depression

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2008-12; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
polysomnography | 4 weeks

SECONDARY OUTCOMES:
Pittsburgh sleep quality index, Heart rate variability, SF-36 | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yen-ying Kung, MD, Principal Investigator — Institute of Traditional Medicine, National Yang-Ming University and Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan